CLINICAL TRIAL: NCT01278888
Title: Minimally Invasive or Open Surgery for Lung Cancer: Pain, Quality of Life and Economics.
Acronym: PLEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter B Licht (Other)
Responsible Party: Sponsor-Investigator, Peter B Licht, Professor, MD, pHd., Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: s-20080085
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Nonsmall Cell Lung Cancer Cellular Diagnosis
Keywords: Lung cancer; Pain; Quality of life; Economy
MeSH Terms: conditions — Lung Neoplasms; Pain | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLEACE 1 (Active Comparator): Anterolateral vs. posterolateral thoracotomy
  Interventions: Procedure: Anterolateral thoracotomy; Procedure: Posterolateral thoracotomy
- PLEACE 2 (Active Comparator): Video assisted thoracic surgery (VATS) vs. anterolateral thoracotomy
  Interventions: Procedure: VATS; Procedure: Anterolateral Thoracotomy

INTERVENTIONS:
Procedure: Anterolateral thoracotomy — Standard anterolateral thoracotomy
  Other Names: ALT
  Arms: PLEACE 1
Procedure: Posterolateral thoracotomy — Standard muscle sparing posterolateral thoracotomy
  Other Names: PLT
  Arms: PLEACE 1
Procedure: VATS — Standard video assisted thoracic surgery, no use of rib-spreader.
  Arms: PLEACE 2
Procedure: Anterolateral Thoracotomy — Standard anterolateral thoracotomy
  Other Names: ALT
  Arms: PLEACE 2

SUMMARY:
Is thoracoscopic surgery better than traditional open surgery for lung cancer?

Video assisted thoracoscopic surgery for lung cancer (VATS) is presumed to be less traumatic than traditional open surgery for lung cancer but this has never been documented in a randomized trial. Some surgeons hesitate to use VATS because it is technically more demanding, others question if the two methods are oncologically equal. Regardless, VATS has been implemented as a routine method for lung cancer surgery several places around the world including Odense University Hospital. The investigators have launched the first randomized controlled trial in the world comparing the two surgical methods to investigate any differences in length of hospitalization, postoperative pain, life quality within the first year, and health economics.

The investigators include patients with stage I and II lung cancer, and randomize between VATS and open surgery in a design where both the patient and doctors doing general rounds in the ward are blinded until discharge because the dressing on the surgical wound is identical, regardless of the surgical method. The surgeon cannot influence clinical decisions including time to discharge, which is decided by other specialist surgeons. Pain evaluation is performed 6 times daily using the VAS-score, life quality is evaluated continuously during the first 12 months using EQ5D and EORTC QLQC-30 questionnaires, and the consumption of analgetics in both groups are monitored via the national prescription database.

Parallel to this trial a similar clinical study, which is also the first of its kind in the world, has been launched for patients with lung cancers not eligible for VATS. They are randomized between the two traditional open surgical methods (anterolateral and posterolateral thoracotomy) - this is also blinded to both patient and doctors doing rounds until discharge from hospital, and endpoint are similar in the two studies.

206 patients have been randomized in the first substudy (VATS vs. open) and 88 in the second substudy (posterolateral vs. anterolateral).

DETAILED DESCRIPTION:
Is minimally invasive surgery for non small cell lung cancer better than traditional open surgery?

Surgical resection remains the best treatment for non small cell lung carcinoma (NSCLC),but unfortunately many patients suffer major postoperative morbidity - pain being the most frequent. It is assumed that newer minimally invasive surgical techniques (Video Assisted Thoracoscopic Surgery - VATS) reduces postoperative morbidity but there is no level 1 evidence available in the literature. This prompted us to perform the present ongoing study, which is the first of its kind in the world.

The investigators compare VATS with traditional open surgery for early stage lung cancer in a clinical randomized double blinded trial. Our aims are to evaluate differences in postoperative pain, life quality, and health economical aspects. The results of this trial could influence future surgical decisionmaking internationally on the surgical treatment for lung cancer.

Likewise, in patients with larger tumours of the lung, which are not suitable for minimally invasive surgery, different techniques are available. The most widely used techniques are the posterolateral thoracotomy and the anterolateral thoracotomy. So far no randomized controlled trail has shown which of these techniques to be superior. This has led us to also randomize between anterolateral and the posterolateral thoracotomy (muscle sparing). The same endpoints are used.

Pain following lung surgery has been a much discussed topic for a long time in the field of thoracic surgery. Depending on the reference, up to 50% of patients develop chronic pain after open lung surgery. Therefore, different surgical approaches have been developed including anterior, lateral or posterior thoracotomy with or without sparing the chest wall muscles. The intercostal nerve is also of concern because of trauma from the rib retractor which is believed to be a cause of both acute and chronic pain. Other concerns are the amount of divided tissue, extend of rib displacement by the rib retractor, type of analgesics, administration form of analgesics, and administration time of the analgesics and it is generally accepted that pain in lung cancer patients is multifactorial.

VATS was introduced in an attempt to reduce the surgical trauma with less tissue damage, avoidance of the rib retraction and the consequently intercostal nerve injury, but never the less several patients develop chronic pain after lung surgery by VATS.

Information on quality of life and health economical aspects following surgery for lung cancer are scarce. No randomized controlled trial has been published. Very little is known if lung cancer patients regain their workability and if so to what extent following surgery.

Likewise, it is not known if VATS is more costly than open procedures, as the opponents say, or if increased expenses during hospitalization are saved by earlier return to work.

End points

1. Postoperative pain evaluated using the VAS-score and the need for prescription analgetics 2, 4, 8, 12, 26 and 52 weeks after surgery.
2. Health related life quality and workability and -efficiency in the same period, using three different questionnaires: two concerning life quality (EORTC-QLQC-30 and EQ5D) and one concerning workability (WPAI).
3. Health economical aspect such as application for pension, visits to general practitioner, readmitted to hospital, number of days away from work due to postoperative morbidity, etc.

All gathered from different databases managed by "Danmarks Statistik" here among the "Landspatientregistret(LPR)", "Sygesikringsstatistikregistret" ,and "Lægemiddelstatistik-registret".

206 patients admitted to the department of cardiothoracic surgery, Odense University Hospital, for elective surgery for lung cancer will be included in each study.

Design

This research project has three sub studies: Two randomized controlled and double blinded clinical trials, and one registry study. One clinical trial randomizes patients with small peripheral lung cancer between VATS (Video Assisted Thoracoscopic Surgery) and standard open anterolateral thoracotomy. The second clinical trial randomizes between anterolateral and posterolateral open thoracotomy in patients not eligible for VATS. The registry sub study monitors patients use of analgetics during the first 12 months (lægemiddelstatestik-registret), their use of other health services, and return to work.

All patients will be operated in general anaesthesia with a double lumen tracheal tube and an epidural catheter. The epidural catheter will be removed when all chest tubes has been removed, but no later than postoperative day 4.

As a standard all patients will be given paracetamol and NSAID in standard doses, and if needed opioids (oxycontin/oxynorm) can be added.

All surgical techniques will be performed as routine operations.

Three different surgical techniques will be used.

1. The VATS approach: one camera port and three assistance ports one of which is enlarged to 5 cm. and rib retractors are never used.
2. Anterolateral thoracotomy: The incision is made from the posterior axillary fold following the linea inframammary to a point below the papilla.
3. Posterolateral thoracotomy. The incision is made from the anterior axillary fold backwards towards the inferior angle of the scapula, without dividing the dorsal latissimus muscle.

In both clinical trials postoperative pain is evaluated by a visual analog scale (VAS). Pain is measured during rest and during coughing. Measurements are done preoperatively and 6 times daily during their hospital stay. After discharge measurements are recorded after 2, 4, 8, 12, 26, and 52 weeks by mail questionnaire.

Both patients and the staff doing general rounds postoperatively will be blinded. In the operating room a dressing will be placed so that it covers the entire hemithorax whereby the incision is hidden. This is done identically regardless of surgical technique. This dressing is left in place until discharge. If changing of the dressing is needed, either the project-nurse or a nurse for another team will assist.

The surgical note is kept in a sealed envelope, which is always placed in the patients chart and can be opened in case of emergency. The chart will only include information about which lobe was resected, no details on the surgical access, but this information is added when the patient is discharged.

The surgeon who has performed the operation will be allowed to check up on their own patients, and to be consulted by the other doctors doing rounds, but they are not allowed to influence on decision-making regarding pain relief or discharge, during the postoperative period.

Timeline

This project is a combination of a ph.d-study and a residency/fellowship in cardiothoracic surgery because this allows for a longer inclusion period. The timeline is divided into three research periods and three clinical periods.

This research project has already been accepted as a ph.d.-project at the University of Southern Denmark, and approved by the local ethical board.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for surgery for lunge cancer.
* Elective surgery (surgery planed > 2 days)
* Accepts randomization
* Age 18 or above.

Exclusion Criteria:

* Previous thoracic surgery
* Planned segment resection or pneumonectomy.
* Any type of chronic pain, requiring daily use of analgetics
* pregnant
* Breast feeding
* T3, T4 tumors or cerebral tumors.
* contraindications to NSAID
* Chemo- and/or radiotherapy in connection to present admission.
* Major surgery planned in connection to this admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2008-09; Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 12 months
  Aim is to asses the development of acute and chronic pain after lobectomy.

SECONDARY OUTCOMES:
Quality of life | 12 months
  Three questionnaires are used. EQ5D, QLQC-30 and WPAI.
Economy | 12 months
  An economical evaluation will be done. Including in-hospital expences, use of sociale-security, readmissions to hospital, use of family practioner, use of and duration of prescription analgetics, wether or not patients are able to return to work, the effect this type of surgery has on the patients quality of life, including a QALY evaluation and cost utility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Licht, Professor, Study Director — Dept. Cardithoracic and Vascular Surgery; Morten Bendixen, MD, Principal Investigator — Dept. Cardiothoracic and Vascular Surgery
Locations (1):
- Odense University Hospital, Odense, Southern Denmark, Denmark

REFERENCES:
- [Derived] Bendixen M, Kronborg C, Jorgensen OD, Andersen C, Licht PB. Cost-utility analysis of minimally invasive surgery for lung cancer: a randomized controlled trial. Eur J Cardiothorac Surg. 2019 Oct 1;56(4):754-761. doi: 10.1093/ejcts/ezz064. PMID 30838382
- [Derived] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473